CLINICAL TRIAL: NCT06507813
Title: A Phase III, Multicenter, Randomized, Double-blind, Controlled Study to Evaluate Pharmacokinetics, Safety and Efficacy of ADC189 Tablets/Granules in Children 2-11 Years Old With Influenza
Brief Title: Safety and Efficacy of ADC189 in Children 2-11 Years Old With Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiaxing AnDiCon Biotech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ADC189GR-20230808
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Influenza Type A; Influenza Type B
MeSH Terms: interventions — baloxavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ADC189 tablets Group (Part 1) (Experimental): Around 30 patients, 6-11 years old.
  Interventions: Drug: ADC189 tablets; Drug: Placebo of Baloxavir Marboxil tablets
- Baloxavir marboxil tablets Group (Part 1) (Active Comparator): Around 15 patients, 6-11 years old.
  Interventions: Drug: Baloxavir Marboxil tablets; Drug: Placebo of ADC189 tablets
- ADC189 granules Group (Part 2A) (Experimental): Around 60 patients, 5-11 years old.
  Interventions: Drug: Placebo of Baloxavir Marboxil tablets; Drug: ADC189 granules
- Baloxavir marboxil tablets (Part 2A) (Active Comparator): Around 30 patients, 5-11 years old.
  Interventions: Drug: Baloxavir Marboxil tablets; Drug: Placebo of ADC189 granules
- ADC189 granules (Part 2B) (Experimental): Around 20 patients, 2-4 years old.
  Interventions: Drug: ADC189 granules; Drug: Placebo of Oseltamivir granules
- Oseltamivir granules (Part 2B) (Active Comparator): Around 10 patients, 2-4 years old.
  Interventions: Drug: Placebo of ADC189 granules; Drug: Oseltamivir granules

INTERVENTIONS:
Drug: ADC189 tablets — Patients weigh between 20 to 80 kilograms, given 45 mg ADC189 tablets once; patients weigh over 80 kilograms, given 90 mg ADC189 tablets once.
  Arms: ADC189 tablets Group (Part 1)
Drug: Baloxavir Marboxil tablets — Patients weigh between 20 to 80 kilograms, given 40 mg Baloxavir marboxil tablets once. Patients weigh over 80 kilograms, given 80 mg Baloxavir marboxil tablets once.
  Arms: Baloxavir marboxil tablets (Part 2A); Baloxavir marboxil tablets Group (Part 1)
Drug: Placebo of ADC189 tablets — Patients weigh between 20 to 80 kilograms, given 1 tablet of placebo once; patients weigh over 80 kilograms, given 2 tablets of placebo once.
  Arms: Baloxavir marboxil tablets Group (Part 1)
Drug: Placebo of Baloxavir Marboxil tablets — Patients weigh between 20 to 80 kilograms, given 2 tablets of placebo once; patients weigh over 80 kilograms, given 4 tablets of placebo once.
  Arms: ADC189 granules Group (Part 2A); ADC189 tablets Group (Part 1)
Drug: ADC189 granules — For patient 5-11 years old, patients weigh between 20 to 80 kilograms, given 45 mg ADC189 granules once; patients weigh over 80 kilograms, given 90 mg ADC189 granules once.
  For patient 2-4 years old, patients <10kg, given 15mg ADC189 granules once. 10kg ~ <15kg, given 25mg ADC189 granules once. 15kg ~<20 kg, given 35mg ADC189 granules once. 20kg ~ <80kg, given 45mg ADC189 granules once.
  Arms: ADC189 granules (Part 2B); ADC189 granules Group (Part 2A)
Drug: Placebo of ADC189 granules — Placebo. Given once only.
  Arms: Baloxavir marboxil tablets (Part 2A); Oseltamivir granules (Part 2B)
Drug: Placebo of Oseltamivir granules — For patients 2-4 years old. Placebo. Given 10 times (5 days, BID).
  Arms: ADC189 granules (Part 2B)
Drug: Oseltamivir granules — For patients 2-4 years old. Patients <15kg, given 30mg×10 times (5 days, BID) Oseltamivir granules. 15kg ~ <23kg, given 45mg×10 times (5 days, BID) Oseltamivir granules. 23kg ~ <40kg, given 60mg×10 times (5 days, BID) Oseltamivir granules. ≥40kg, given 75mg×10 times (5 days, BID) Oseltamivir granules.
  Arms: Oseltamivir granules (Part 2B)

SUMMARY:
Currently, there is only one treatment which only need one single oral dose for influenza in children five years above (Baloxavir marboxil) in China. This study will test a medicine for influenza in children younger than 5 year of age to see if it is safe and effective.

This is a multicenter, randomized, double-blind, controlled Phase III clinical study.

The study evaluates the pharmacokinetics, safety and efficacy of ADC189 tablets/granules following a single oral dose in children aged 2 to 11 years with influenza.

ELIGIBILITY:
Key Inclusion Criteria:

* 1. Patients aged 2 to 11 years at screening, both sex;
* 2. Patients were diagnosed with Influenza A Vairus Infection/Influenza B Virus Infection.
* 3. Parents willing and able to comply with study requirements, under the judgment of investigators .
* 4. Onset of symptoms no more than 48 hours before presentation for screening.

Key Exclusion Criteria:

* 1. Patients with severe influenza.
* 2. Pregnant or breast-feeding females
* 3. Patients with acute respiratory infection, tympanitis, sinusitis, or acute asthma attack within 2 weeks before screening.
* 4. Presence of a chronic disease or illness that may indicate increased risk for influenza-related complications.
* 5. Other antiviral therapy is required during screening.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
The safety of study drug, Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to 15 days
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/ incapacity, is a congenital anomaly/ birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above.

SECONDARY OUTCOMES:
Plasma Concentrations of ADC189 and ADC189-I07 | From Day 1 up to 14 days, 4 time points.
  ADC189-I07 is an active metabolite of ADC189. Four plasma samples were collected in 4 time points from each patient. This data is collected for Pop PK analysis.
Time to Resolution of Influenza Symptoms | From Day 1 up to 14 days
  Subjects or parents or caregivers were asked to provide an assessment of age-appropriate influenza symptoms on a CARIFS Questionare.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No